CLINICAL TRIAL: NCT02819232
Title: Microbiological Diagnosis of Infectious Keratitis to Pathogenic Fastidious Germs
Acronym: Keratite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-40; 2012-A01568-35 (Other: ANSM)
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Infectious Keratitis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with a prescription of a microbiologic diagnostic of (Other): Patient with a prescription of a microbiologic diagnostic of keratitis
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Detection of bacteria will be performed on a blood sample

SUMMARY:
Infectious keratitis are favored by the circumstances causing the small trauma of the corneal epithelium, corneal surgery, corneal dryness under health system such as Sjögren's syndrome rheumatoid arthritis, or much more frequently wearing contact lenses. If the majority of infectious keratitis are favourable, some lead to serious injury of the cornea, or even corneal perforation which result an endophthalmitis. This unfavourable evolution may lead to blindness due to corneal damage, the endo-ocular lesions or enucleation of the eyeball. This negative evolution is encountered while the infectious keratitis due to tedious germs of difficult diagnosis such as nontuberculous Mycobacterial, fungal infections, fungal keratitis, amoebic keratitis, and certain viral keratitis. The microbiological diagnosis of routine is based on the systematic search for pathogens tedious from invasive sampling of cornea by vaccinostyle. We set up a new non-invasive corneal swab diagnostic method.

DETAILED DESCRIPTION:
Primary Purpose: Compare the ability diagnostic of non-invasive sampling swab corneal versus the gold standard, (invasive vaccinostyle uptake) for the systematic search for pathogens tedious in corneal specimens.

Hypothesis:

The diagnostic strategy using a microbial testing of cornea method has a sensitivity of 90% and a specificity of 80% or more over the policy diagnostic using a sampling by vaccinostyle method.

Primary outcome measures: Sensitivity, specificity, positive and negative predictive values, Diagnostic odds ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patient is more than 18 years old.
* Patient with a prescription of a microbiologic diagnostic of keratitis
* Patient who do not declined to have his medical records reviewed for research
* Patient with health insurance

Exclusion Criteria:

* minor patient (<18 years).
* Pregnant or breastfeeding women.
* Major Patient under guardianship.
* Patient in vital emergency.
* Private Patient liberty or under court order.
* Patient refusing to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2013-08-12 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive and negative predictive values, Diagnostic odds ratio. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Michel Drancourt, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided